CLINICAL TRIAL: NCT00543244
Title: Early Prediction of Successful Treatment for Chronic Hepatitis C Virus Infection in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200709053R
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-02

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Pegylated interferon; Ribavirin; Virokinetics
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients with chronic hepatitis C who receive pegylated interferon plus ribavirin for 24 weeks (genotype 1 or 2) and for 48 weeks (genotype 1)
  Interventions: Drug: Pegylated interferon alfa and ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa and ribavirin — Pegylated interferon alfa-2a 180 ug/week or pegylated interferon alfa-2b 1.5 ug/kg/week Ribavrin 800-1200 mg/day (genotype 1: < 75 kg 1000 mg/day, >=75 kg 1200 mg/day; genotype 2: 800 mg/day)
  HCV genotype: baseline (Day 0) HCV RNA (real time PCR test): baseline (Day 0), Day 1 (4,8,12 hours after pegylated interferon + ribavirin), Day 2 (24,36 hours), Day 3(48 hours), Day 4 (72 hours), Day 5 (96 hours), Week 2,4,6,8,12,16,20,24, and 28,32,36,40,44,48,72 (for genotype 1 with 48 weeks of treatment), and 48 (for genotype 1 or 2 with 24 weeks of treatment)
  Other Names: Pegasys plus Robatrol; Peg-Intron plus Rebetol

SUMMARY:
Hepatitis C virus (HCV) infection is a global health problem, which may lead to chronic hepatitis, cirrhosis, hepatic decompensation and hepatocellular carcinoma (HCC). Recently, treatment with peginterferon alfa plus ribavirin has become the standard of care for patients with chronic hepatitis C. While genotype 2 patients can have higher sustained virologic response (SVR) rates to 80-90%, genotype 1 patients generally have low SVR rates of only 40-50%. In contrast, genotype 1 Taiwanese patients have superior SVR rates than those in Western countries. Despite the overall improved response to this combination therapy, more than 75% of patients suffer from treatment-related adverse events and the costs remain high, which make individualized therapy of paramount importance to maximize treatment response and minimize adverse events.

HCV viral kinetics with interferon-based therapies have been studied recently to evaluate patient responses. Early viral kinetics shown to have favorable SVR rates, which make shorter treatment duration possible. However, different viral kinetics were found through ethnicity. Recently, a pilot study to evaluate the viral kinetics of 6 Taiwanese patients with HCV infection who received peginterferon alfa plus ribavirin therapy has shown superior early viral kinetics to those in Caucasian patients. Based on the favorable SVR rates in treating Taiwanese patients with chronic hepatitis C, the investigators aimed to conduct a large confirmatory study to evaluate the viral kinetics and try to define the optimal treatment for these patients.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a global health problem, which may lead to chronic hepatitis, cirrhosis, hepatic decompensation and hepatocellular carcinoma (HCC). [1,2] Recently, treatment with peginterferon alfa plus ribavirin has become the standard of care for patients with chronic hepatitis C. While genotype 2 patients can have higher sustained virologic response (SVR) rates to 80-90%, genotype 1 patients generally have low SVR rates of only 40-50%. [3-5] In contrast, genotype 1 Taiwanese patients have superior SVR rates that those in Western countries. [6,7] Despite the overall improved response to this combination therapy, more than 75% of patients suffer from treatment-related adverse events and the costs remain high, [8,9] which make individualized therapy of paramount importance to maximize treatment response and minimize adverse events.

HCV viral kinetics with interferon-based therapies have been studied recently to evaluate patient responses. [10-14] Early viral kinetics shown to have favorable SVR rates, which make shorter treatment duration possible. [15-18] However, different viral kinetics were found through ethnicity. [19-23] Recently, a pilot study to evaluate the viral kinetics of 6 Taiwanese patients with HCV infection who received peginterferon alfa plus ribavirin therapy has shown superior early viral kinetics to those in Caucasian patients. [24] Based on the favorable SVR rates in treating Taiwanese patients with chronic hepatitis C, the investigators aimed to conduct a large confirmatory study to evaluate the viral kinetics and try to define the optimal treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* Over 18 years old
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Amplicor HCV Monitor v2.0, Roche Molecular Systems, Pleasanton, CA) with dynamic range 600~< 500,000 IU/ml
* Serum alanine aminotransferase levels above the upper limit of normal with 6 months of enrollment
* A liver biopsy consistent with the diagnosis of chronic hepatitis C

Exclusion Criteria:

* Anemia (hemoglobin < 13 gram per deciliter for men and < 12 gram per deciliter for women)
* Neutropenia (neutrophil count < 1,500 per cubic milliliter)
* Thrombocytopenia (platelet < 90,000 per cubic milliliter)
* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Chronic alcohol abuse (daily consumption > 20 gram per day)
* Decompensated liver disease (Child-Pugh class B or C)
* Serum creatinine level more than 1.5 times the upper limit of normal
* Autoimmune liver disease
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception
* Unwilling to receive serial blood sampling during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C virus infection who receive pegylated interferon plus ribavirin for an overall of 24-48 weeks
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-10 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 1~1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, MD, PhD, Study Chair — National Taiwan University Hospital; Avidan Uriel Neumann, PhD, Principal Investigator — Faculty of Life Sciences, Bar-Ilan University, Ramat-Gan, Israel; Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (7):
- Faculty of Life Sciences, Bar-Ilan University, Ramat Gan, Israel
- Taiwan (6):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Buddhist Tzu Chi General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Ren-Ai Branch, Taipei Municipal Hospital, Taipei

REFERENCES:
- [Background] Chen DS, Kuo GC, Sung JL, Lai MY, Sheu JC, Chen PJ, Yang PM, Hsu HM, Chang MH, Chen CJ, et al. Hepatitis C virus infection in an area hyperendemic for hepatitis B and chronic liver disease: the Taiwan experience. J Infect Dis. 1990 Oct;162(4):817-22. doi: 10.1093/infdis/162.4.817. PMID 2169497
- [Background] Lai MY. Combined interferon and ribavirin therapy for chronic hepatitis C in Taiwan. Intervirology. 2006;49(1-2):91-5. doi: 10.1159/000087269. PMID 16166795
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Hadziyannis SJ, Sette H Jr, Morgan TR, Balan V, Diago M, Marcellin P, Ramadori G, Bodenheimer H Jr, Bernstein D, Rizzetto M, Zeuzem S, Pockros PJ, Lin A, Ackrill AM; PEGASYS International Study Group. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004 Mar 2;140(5):346-55. doi: 10.7326/0003-4819-140-5-200403020-00010. PMID 14996676
- [Background] Lee SD, Yu ML, Cheng PN, Lai MY, Chao YC, Hwang SJ, Chang WY, Chang TT, Hsieh TY, Liu CJ, Chen DS. Comparison of a 6-month course peginterferon alpha-2b plus ribavirin and interferon alpha-2b plus ribavirin in treating Chinese patients with chronic hepatitis C in Taiwan. J Viral Hepat. 2005 May;12(3):283-91. doi: 10.1111/j.1365-2893.2005.00590.x. PMID 15850469
- [Background] Yu ML, Dai CY, Lin ZY, Lee LP, Hou NJ, Hsieh MY, Chen SC, Hsieh MY, Wang LY, Chang WY, Chuang WL. A randomized trial of 24- vs. 48-week courses of PEG interferon alpha-2b plus ribavirin for genotype-1b-infected chronic hepatitis C patients: a pilot study in Taiwan. Liver Int. 2006 Feb;26(1):73-81. doi: 10.1111/j.1478-3231.2005.01196.x. PMID 16420512
- [Background] Strader DB, Wright T, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C. Hepatology. 2004 Apr;39(4):1147-71. doi: 10.1002/hep.20119. No abstract available. PMID 15057920
- [Background] Fried MW. Side effects of therapy of hepatitis C and their management. Hepatology. 2002 Nov;36(5 Suppl 1):S237-44. doi: 10.1053/jhep.2002.36810. PMID 12407599
- [Background] Neumann AU, Lam NP, Dahari H, Gretch DR, Wiley TE, Layden TJ, Perelson AS. Hepatitis C viral dynamics in vivo and the antiviral efficacy of interferon-alpha therapy. Science. 1998 Oct 2;282(5386):103-7. doi: 10.1126/science.282.5386.103. PMID 9756471
- [Background] Lee WM, Reddy KR, Tong MJ, Black M, van Leeuwen DJ, Hollinger FB, Mullen KD, Pimstone N, Albert D, Gardner S. Early hepatitis C virus-RNA responses predict interferon treatment outcomes in chronic hepatitis C. The Consensus Interferon Study Group. Hepatology. 1998 Nov;28(5):1411-5. doi: 10.1002/hep.510280533. PMID 9794929
- [Background] Orito E, Mizokami M, Suzuki K, Ohba K, Ohno T, Mori M, Hayashi K, Kato K, Iino S, Lau JY. Loss of serum HCV RNA at week 4 of interferon-alpha therapy is associated with more favorable long-term response in patients with chronic hepatitis C. J Med Virol. 1995 Jun;46(2):109-15. doi: 10.1002/jmv.1890460205. PMID 7636496
- [Background] Colombatto P, Civitano L, Oliveri F, Coco B, Ciccorossi P, Flichman D, Campa M, Bonino F, Brunetto MR. Sustained response to interferon-ribavirin combination therapy predicted by a model of hepatitis C virus dynamics using both HCV RNA and alanine aminotransferase. Antivir Ther. 2003 Dec;8(6):519-30. PMID 14760885
- [Background] Herrmann E, Lee JH, Marinos G, Modi M, Zeuzem S. Effect of ribavirin on hepatitis C viral kinetics in patients treated with pegylated interferon. Hepatology. 2003 Jun;37(6):1351-8. doi: 10.1053/jhep.2003.50218. PMID 12774014
- [Background] Jessner W, Stauber R, Hackl F, Datz C, Watkins-Riedel T, Hofer H, Gangl A, Kessler H, Ferenci P. Early viral kinetics on treatment with pegylated interferon-alpha-2a in chronic hepatitis C virus genotype 1 infection. J Viral Hepat. 2003 Jan;10(1):37-42. doi: 10.1046/j.1365-2893.2003.00396.x. PMID 12558910
- [Background] Carlsson T, Reichard O, Norkrans G, Blackberg J, Sangfelt P, Wallmark E, Weiland O. Hepatitis C virus RNA kinetics during the initial 12 weeks treatment with pegylated interferon-alpha 2a and ribavirin according to virological response. J Viral Hepat. 2005 Sep;12(5):473-80. doi: 10.1111/j.1365-2893.2005.00621.x. PMID 16108761
- [Background] Ouzan D, Khiri H, Penaranda G, Joly H, Halfon P. Kinetics of hepatitis C virus RNA load during pegylated interferon alpha-2a and ribavirin treatment in naive genotype 1 patients. Comp Hepatol. 2005 Dec 21;4:9. doi: 10.1186/1476-5926-4-9. PMID 16371151
- [Background] Jensen DM, Morgan TR, Marcellin P, Pockros PJ, Reddy KR, Hadziyannis SJ, Ferenci P, Ackrill AM, Willems B. Early identification of HCV genotype 1 patients responding to 24 weeks peginterferon alpha-2a (40 kd)/ribavirin therapy. Hepatology. 2006 May;43(5):954-60. doi: 10.1002/hep.21159. PMID 16628671
- [Background] Reddy KR, Hoofnagle JH, Tong MJ, Lee WM, Pockros P, Heathcote EJ, Albert D, Joh T. Racial differences in responses to therapy with interferon in chronic hepatitis C. Consensus Interferon Study Group. Hepatology. 1999 Sep;30(3):787-93. doi: 10.1002/hep.510300319. PMID 10462387
- [Background] McHutchison JG, Poynard T, Pianko S, Gordon SC, Reid AE, Dienstag J, Morgan T, Yao R, Albrecht J. The impact of interferon plus ribavirin on response to therapy in black patients with chronic hepatitis C. The International Hepatitis Interventional Therapy Group. Gastroenterology. 2000 Nov;119(5):1317-23. doi: 10.1053/gast.2000.19289. PMID 11054390
- [Background] Layden-Almer JE, Ribeiro RM, Wiley T, Perelson AS, Layden TJ. Viral dynamics and response differences in HCV-infected African American and white patients treated with IFN and ribavirin. Hepatology. 2003 Jun;37(6):1343-50. doi: 10.1053/jhep.2003.50217. PMID 12774013
- [Background] Hepburn MJ, Hepburn LM, Cantu NS, Lapeer MG, Lawitz EJ. Differences in treatment outcome for hepatitis C among ethnic groups. Am J Med. 2004 Aug 1;117(3):163-8. doi: 10.1016/j.amjmed.2004.02.043. PMID 15276594
- [Background] Yu ML, Chuang WL, Dai CY, Lee LP, Hsieh MY, Lin ZY, Chen SC, Hsieh MY, Wang LY, Chang WY, Tsai SL, Kuo HT. Different viral kinetics between hepatitis C virus genotype 1 and 2 as on-treatment predictors of response to a 24-week course of high-dose interferon-alpha plus ribavirin combination therapy. Transl Res. 2006 Sep;148(3):120-7. doi: 10.1016/j.trsl.2006.04.006. PMID 16938649
- [Background] Hsu CS, Liu CJ, Lai MY, Chen PJ, Kao JH, Chen DS. Early viral kinetics during treatment of chronic hepatitis C virus infection with pegylated interferon alpha plus ribavirin in Taiwan. Intervirology. 2007;50(4):310-5. doi: 10.1159/000105444. Epub 2007 Jul 9. PMID 17622791